CLINICAL TRIAL: NCT03718325
Title: Clinical Characterization of Burst Spinal Cord Stimulation for Chronic Pain Management
Brief Title: Burst Spinal Cord Stimulation (Burst-SCS) Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated early due to data quality concerns and protocol integrity issues involving inadequate sham stimulation parameters and compromised participant blinding.
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Scott Lempka, Associate Professor of Biomedical Engineering and Associate Professor of Anesthesiology, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00147961; UL1TR002240 (NIH)
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Results first posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Pain, Chronic; Failed Back Surgery Syndrome
Keywords: Burst-SCS; Chronic pain; Spinal cord stimulation
MeSH Terms: conditions — Chronic Pain; Failed Back Surgery Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: There will be two research teams. One team will be unblinded (e.g. clinical care provider/company representative, study coordinator) and will perform stimulator programming/adjustment, and the other team will be blinded (e.g. research personnel) and will perform clinical testing and collect study outcome measures.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Burst-SCS/sham SCS (Other): First, participants will receive Burst-SCS. Study evaluations will be completed prior to and after stimulation. Then, participants will have their stimulation adjusted to receive sham (no) SCS. Study evaluations will be completed prior to and after this sham.
  Interventions: Device: Burst-SCS; Device: Sham SCS
- Sham SCS/Burst-SCS (Other): First, participants will receive sham (no) SCS. Study evaluations will be completed prior to and after this sham. Then, participants will have their stimulation adjusted to receive Burst-SCS. Study evaluations will be completed prior to and after stimulation.
  Interventions: Device: Burst-SCS; Device: Sham SCS

INTERVENTIONS:
Device: Burst-SCS — The treatment arm used in the study is burst spinal cord stimulation (Burst-SCS). The device used to deliver Burst-SCS is the St. Jude Medical Invisible Trial System.
Device: Sham SCS — The placebo control arm used in the study is sham spinal cord stimulation (sham SCS). The device used to deliver sham SCS is the St. Jude Medical Invisible Trial System.

SUMMARY:
Recently a new form of spinal cord stimulation therapy called burst spinal cord stimulation (Burst-SCS) is available to treat chronic pain. The goal of this study is to learn more about how Burst-SCS works to reduce chronic pain. The study will examine chronic pain patients who have been deemed candidates for Burst-SCS therapy, and who have already been selected to receive a temporary externalized trial of Burst-SCS from their own doctors as part of their standard clinical care for chronic pain management. During the study, participants will be asked to complete a variety of evaluations at certain time points. In addition, there will be a randomized, double blind, crossover phase, where the particular effects of Burst-SCS and sham SCS will be evaluated. The device used to deliver Burst-SCS and sham SCS is the St. Jude Medical Invisible Trial System.

DETAILED DESCRIPTION:
The study was terminated early following the identification of data quality concerns and protocol integrity issues, specifically related to inadequate sham stimulation parameters and compromised participant blinding. Results reporting was significantly delayed due to research-related pauses during the COVID-19 pandemic. Although there were initial plans to resume enrollment and study procedures once feasible, a comprehensive review of the study data identified the protocol integrity concerns, leading to the decision to terminate the study.

ELIGIBILITY:
Inclusion Criteria:

* Men or women with chronic, intractable pain of the trunk and/or limbs, including unilateral or bilateral pain associated with any of the following: failed back surgery syndrome and intractable low back and leg pain, and for whom Burst-SCS has been recommended as a treatment option
* Candidates who can speak, read, and understand English

Exclusion Criteria:

* Subjects who are pregnant- as determined by verbal report or chart review
* Subjects with current, habitual, or previous use within the last 12 months of artificial nails, nail enhancements, or nail extensions that cover any portion of either thumbnail. Exceptions, including brief and/or occasional use, may be permissible at the discretion of the principal investigator
* Subjects who are unable or unwilling to cooperate with clinical testing
* Subjects having any impairment, activity or situation that, in the judgement of the study coordinator or PI, would prevent satisfactory completion of the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Lempka, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twelve participants were enrolled and had baseline data collected, with nine proceeding to randomization. There were no washout periods between points of data collection during the crossover phase of the trial.
Groups:
- Un-randomized Participants: Participants who were evaluated at baseline but did not undergo randomization. Un-randomized participants did not receive any SCS as part of the research study.
- Burst-SCS/Sham-SCS: First, participants will receive Burst-SCS. Study evaluations will be completed prior to and after stimulation. Then, participants will have their stimulation adjusted to receive sham (no) SCS. Study evaluations will be completed prior to and after this sham.
  Burst-SCS: The treatment arm used in the study is burst spinal cord stimulation (Burst-SCS). The device used to deliver Burst-SCS is the St. Jude Medical Invisible Trial System.
  Sham SCS: The placebo control arm used in the study is sham spinal cord stimulation (sham SCS). The device used to deliver sham SCS is the St. Jude Medical Invisible Trial System.
- Sham-SCS/Burst-SCS: First, participants will receive sham (no) SCS. Study evaluations will be completed prior to and after this sham. Then, participants will have their stimulation adjusted to receive Burst-SCS. Study evaluations will be completed prior to and after stimulation.
  Burst-SCS: The treatment arm used in the study is burst spinal cord stimulation (Burst-SCS). The device used to deliver Burst-SCS is the St. Jude Medical Invisible Trial System.
  Sham SCS: The placebo control arm used in the study is sham spinal cord stimulation (sham SCS). The device used to deliver sham SCS is the St. Jude Medical Invisible Trial System.
Period: Overall Study
Arm/Group | Un-randomized Participants | Burst-SCS/Sham-SCS | Sham-SCS/Burst-SCS
Started (Baseline visit) | 3 | 4 | 5
Period 1 (up to 28 Days After Baseline Visit) | 0 | 4 | 5
Period 2 (up to 1 Day After Period 1 Visit) | 0 | 4 | 5
Completed | 0 | 4 | 5
Not Completed | 3 | 0 | 0
Not completed — Externalized leads were removed independent of the research protocol | 2 | 0 | 0
Not completed — Lost to follow-up because of research pause caused by the COVID-19 pandemic | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Burst-SCS/Sham-SCS | Sham-SCS/Burst-SCS | Un-randomized Participants | Total
Number analyzed (Participants) | 4 | 5 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (10.1) | 51.8 (8.64) | 48.7 (6.81) | 50.6 (8.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 6
  Male | 1 | 3 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 5 | 3 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 5 | 3 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 5 | 3 | 12
Visual Analog Scale (VAS) Score [Mean (Standard Deviation); unit: score on a scale] — VAS was a horizontal line 100 millimeters (mm) in length with the word "no pain" and "worst possible pain" printed below. The participant marked on the line the point that they felt represented their perception of their current state. The score was determined by measuring in millimeters from the left hand with a total range of 0-100 millimeters, with a score between 0 (no pain) to a score of 100 (worst possible pain). Higher VAS values represented more severe pain and lower values represented lower pain.
  score on a scale | 71.2 (9.60) | 78.4 (15.0) | 83.7 (5.20) | 76.8 (12.0)
Short-Form McGill Pain Questionnaire (SFMPQ) Score [Mean (Standard Deviation); unit: score on a scale] — SFMPQ was used to describe the quality of pain and had 15 descriptors (11 sensory and 4 affective). Each descriptor was scored by a 4-point intensity scale (0=none to 3=severe) (range 0-45). Pain scores were derived from the sum of the intensity rank values of the words chosen for sensory, affective, and total descriptors.
  score on a scale | 26 (11.2) | 19.6 (10.7) | 22.7 (1.53) | 22.5 (9.20)
General Pain Disability Index (PDI) Score [Mean (Standard Deviation); unit: score on a scale] — Pain-related disability was assessed using the six-item General Pain Disability Index Questionnaire, which measures the degree to which chronic pain disrupts various aspects of daily life. Each item is rated on a 0-10 scale where 0 indicates no disability and 10 indicates total disability in that activity due to pain. The total score ranges from 0 to 60, with higher scores indicating greater pain-related disability.
  score on a scale | 36.3 (5.62) | 30.6 (11.9) | 24.7 (17.0) | 31 (11.6)
Brief Pain Inventory-Short Form (BPI-SF) Score [Mean (Standard Deviation); unit: score on a scale] — Pain severity and interference were assessed using the Brief Pain Inventory (BPI). The instrument includes four items measuring pain severity and seven items measuring pain interference with daily activities. Each item is rated on a 0-10 numerical rating scale. A total composite BPI-SF score was calculated by summing severity (range 0-40) and interference (range 0-70) domains for a total score of 0-110. Higher scores indicate greater pain burden and impairment.
  score on a scale | 6.84 (0.71) | 6.59 (2.19) | 6.12 (1.36) | 6.56 (1.52)
Michigan Body Map (MBM) [Mean (Standard Deviation); unit: checked boxes] — MBM was used to assess body areas where chronic pain was experienced and quantify the degree of widespread body pain (i.e. pain centralization). Pain spread was collected by having participants check all areas of the body as outlined on the body map where they felt persistent or recurrent pain. A checked box meant pain was present in that region of the body. The MBM had 35 boxes total participants could check, which were summed together to assess participants' pain. Lower number of checked boxes indicated less widespread pain; higher number of checked boxes indicated more widespread pain.
  checked boxes | 4.5 (5.69) | 7.2 (5.45) | 11.3 (7.77) | 7.33 (6.14)
Fibromyalgia Survey Questionnaire (FSQ) - Widespread Pain Index [Mean (Standard Deviation); unit: score on a scale] — Pain distribution was assessed using the Widespread Pain Index (WPI) component of the Fibromyalgia Survey Questionnaire (FSQ). The WPI is a 19-item checklist that evaluates the presence of pain or tenderness in 19 specific body regions. Each painful area receives a score of 1, with the total WPI score ranging from 0 to 19, where higher scores indicate more widespread pain distribution.
  score on a scale | 3.25 (3.86) | 3.8 (2.05) | 5.67 (2.52) | 4.08 (2.78)
Fibromyalgia Survey Questionnaire (FSQ) - Symptom Severity Index [Mean (Standard Deviation); unit: score on a scale] — The Symptom Severity Index (SSI) component of the FSQ includes two sections: (1) a 3-item scale assessing fatigue, cognitive symptoms, and waking unrefreshed, each rated on a 0-3 scale (0=no problem, 1=mild, 2=moderate, 3=severe); and (2) a 3-item checklist evaluating the presence of lower abdominal pain, depression, and headache (0=absent, 1=present). Total scores range from 0 to 12, with higher scores indicating greater symptom severity.
  score on a scale | 7.00 (2.16) | 3.20 (1.92) | 5.67 (0.58) | 5.08 (2.39)

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analog Scale (VAS) Score
Description: Visual analog scale (VAS) was a horizontal line 100 millimeters (mm) in length with the word "no pain" and "worst possible pain" printed below. The participant marked on the line the point that they felt represented their perception of their current state. The score was determined by measuring in millimeters from the left hand with a total range of 0-100 millimeters, with a score between 0 (no pain) to a score of 100 (worst possible pain). Higher VAS values represented more severe pain and lower values represented lower pain. Change from baseline scores are calculated as the follow-up score minus the baseline score, where negative values indicate improvement (reduced pain) and positive values indicate worsening (increased pain). Results were aggregated from all interventions regardless of treatment order and reflect the total difference from baseline.
Time Frame: Up to one month following the pre-implant visit.
Population: Of the 9 randomized participants, usable data was only obtained from 3 participants due to protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Change of Burst-SCS From Pre-implant: Burst-SCS: The treatment arm used in the study is burst spinal cord stimulation (Burst-SCS). The device used to deliver Burst-SCS is the St. Jude Medical Invisible Trial System.
  Pre-implant: Pre-operative baseline assessment prior to implantation of the spinal cord stimulation (SCS) electrode arrays.
- Change of Sham-SCS From Pre-implant: Sham SCS: The placebo control arm used in the study is sham spinal cord stimulation (sham SCS). The device used to deliver sham SCS is the St. Jude Medical Invisible Trial System.
  Pre-implant: Pre-operative baseline assessment prior to implantation of the spinal cord stimulation (SCS) electrode arrays.
Arm/Group | Change of Burst-SCS From Pre-implant | Change of Sham-SCS From Pre-implant
Number analyzed (Participants) | 3 | 3
score on a scale
  Baseline - Usable Data | 81.1 (20.1) | 81.1 (20.1)
  Change - Usable Data | -44.7 (47.9) | -44.7 (49.6)

2. Secondary Outcome: Change in Short-Form McGill Pain Questionnaire (SFMPQ) Score
Description: The Short-Form McGill Pain Questionnaire (SFMPQ) assesses the quality and intensity of pain using 15 descriptors representing sensory (11 items) and affective (4 items) dimensions of pain. Each descriptor is rated on a 4-point intensity scale where 0=none, 1=mild, 2=moderate, and 3=severe. The total scores are calculated by summing the intensity ratings for each of the 15 descriptors (possible score range 0 to 45). Higher scores indicate more severe pain symptoms. Change from baseline scores are calculated as the follow-up score minus the baseline score, where negative values indicate improvement (reduced pain; better outcome) and positive values indicate worsening (increased pain; worse outcome). Results were aggregated from all interventions regardless of treatment order and reflect the total difference from baseline.
Time Frame: Up to one month following the pre-implant visit.
Population: Of the 9 randomized participants, usable data was only obtained from 3 participants due to protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Change of Burst-SCS From Pre-implant | Change of Sham-SCS From Pre-implant
Number analyzed (Participants) | 3 | 3
score on a scale
  Baseline - Usable Data | 17.7 (9.81) | 17.7 (9.81)
  Change - Usable Data | -11.67 (9.50) | -7.67 (7.51)

3. Secondary Outcome: Change in General Pain Disability Index (PDI) Score
Description: Pain-related disability was assessed using the six-item General Pain Disability Index (PDI) Questionnaire, which measures the degree to which chronic pain disrupts various aspects of daily life. Each item is rated on a 0-10 scale where 0 indicates no disability and 10 indicates total disability in that activity due to pain. The total score ranges from 0 to 60, with higher scores indicating greater pain-related disability. Change from baseline scores are calculated as the follow-up score minus the baseline score, where negative values indicate improvement (reduced pain-disability) and positive values indicate worsening (increased pain-related disability). Results were aggregated from all interventions regardless of treatment order and reflect the total difference from baseline.
Time Frame: Up to one month following the pre-implant visit.
Population: Of the 9 randomized participants, usable data was only obtained from 3 participants due to protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Change of Burst-SCS From Pre-implant | Change of Sham-SCS From Pre-implant
Number analyzed (Participants) | 3 | 3
score on a scale
  Baseline - Usable Data | 38.3 (9.02) | 38.3 (9.02)
  Change - Usable Data | -19.00 (24.76) | -20.33 (24.79)

4. Secondary Outcome: Change in Brief Pain Inventory-Short Form (BPI-SF) Score
Description: The Brief Pain Inventory-Short Form (BPI-SF) assesses pain severity and pain interference with daily functioning. It includes four items assessing pain severity (worst, least, average, current) and seven items assessing interference (general activity, mood, walking, work, relations, sleep, enjoyment of life). Each item is rated 0 (no pain/interference) to 10 (worst pain/interferes completely). A total composite BPI-SF score was calculated by summing severity (range 0-40) and interference (range 0-70) domains for a total score of 0-110. Higher scores indicate greater pain burden and impairment. Change from baseline was calculated as follow-up score minus baseline score, where negative values indicate improvement. Results were aggregated from all interventions regardless of treatment order and reflect the total difference from baseline.
Time Frame: Up to one month following the pre-implant visit.
Population: Of the 9 randomized participants, usable data was only obtained from 3 participants due to protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Change of Burst-SCS From Pre-implant | Change of Sham-SCS From Pre-implant
Number analyzed (Participants) | 3 | 3
score on a scale
  Baseline - Usable Data | 7.52 (2.15) | 7.52 (2.15)
  Change - Usable Data | -4.12 (5.11) | -3.94 (5.28)

5. Secondary Outcome: Michigan Body Map (MBM)
Description: MBM was used to assess body areas where chronic pain was experienced and quantify the degree of widespread body pain (i.e. pain centralization). Pain spread was collected by having participants check all areas of the body as outlined on the body map where they felt persistent or recurrent pain. A checked box meant pain was present in that region of the body. The MBM had 35 boxes total participants could check, which were summed together to assess participants' pain. Lower number of checked boxes indicated less widespread pain; higher number of checked boxes indicated more widespread pain. Change from baseline scores are calculated as the follow-up score minus the baseline score, where negative values indicate improvement (reduced pain areas) and positive values indicate worsening (increased pain areas). Results were aggregated from all interventions regardless of treatment order and reflect the total difference from baseline.
Time Frame: Up to one month following the pre-implant visit.
Population: Of the 9 randomized participants, usable data was only obtained from 3 participants due to protocol deviations.
Measure: Mean (Standard Deviation); unit: checked boxes
Arm/Group | Change of Burst-SCS From Pre-implant | Change of Sham-SCS From Pre-implant
Number analyzed (Participants) | 3 | 3
checked boxes
  Baseline - Usable Data | 6.67 (8.08) | 6.67 (8.08)
  Change - Usable Data | -5.33 (9.24) | -5.33 (9.24)

6. Secondary Outcome: Fibromyalgia Survey Questionnaire (FSQ) - Widespread Pain Index
Description: Pain distribution was assessed using the Widespread Pain Index (WPI) component of the Fibromyalgia Survey Questionnaire (FSQ). The WPI is a 19-item checklist that evaluates the presence of pain or tenderness in specific body regions experienced during the past 7 days. Participants indicate whether they experienced pain in each of 19 anatomical areas including: bilateral shoulder, upper arm, lower arm, hip, upper leg, lower leg, and jaw; plus neck, upper back, lower back, chest, and abdomen. Each painful area receives a score of 1, with the total WPI score ranging from 0 to 19, where higher scores indicate more widespread pain distribution. Change from baseline scores are calculated as the follow-up score minus the baseline score, where negative values indicate improvement (reduced pain areas) and positive values indicate worsening (increased pain areas). Results were aggregated from all interventions regardless of treatment order and reflect the total diff
Time Frame: Up to one month following the pre-implant visit.
Population: Of the 9 randomized participants, usable data was only obtained from 3 participants due to protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Change of Burst-SCS From Pre-implant | Change of Sham-SCS From Pre-implant
Number analyzed (Participants) | 3 | 3
score on a scale
  Baseline - Usable Data | 3.00 (2.65) | 3.00 (2.65)
  Change - Usable Data | -2.67 (2.89) | -2.00 (3.46)

7. Secondary Outcome: Fibromyalgia Survey Questionnaire (FSQ) - Symptom Severity Index
Description: Symptom severity was assessed using the Symptom Severity Index component of the Fibromyalgia Survey Questionnaire (FSQ). The Symptom Severity Index evaluates fibromyalgia-related symptoms through two sections: (1) a three-item scale assessing fatigue, trouble thinking or remembering, and waking up tired over the past week, each rated on a 0-3 scale (0 = no problem, 1 = slight/mild, 2 = moderate, 3 = severe); and (2) a three-item checklist evaluating the presence of lower abdominal pain/cramps, depression, and headache over the past 6 months (0 = absent, 1 = present). The total Symptom Severity Index score ranges from 0 to 12, with higher scores indicating greater symptom severity. Change from baseline scores are calculated as the follow-up score minus the baseline score, where negative values indicate improvement and positive values indicate worsening. Results were aggregated from all interventions regardless of treatment order and reflect the total difference from baseline.
Time Frame: Up to one month following the pre-implant visit.
Population: Of the 9 randomized participants, usable data was only obtained from 3 participants due to protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Change of Burst-SCS From Pre-implant | Change of Sham-SCS From Pre-implant
Number analyzed (Participants) | 3 | 3
score on a scale
  Baseline - Usable Data | 3.67 (3.21) | 3.67 (3.21)
  Change - Usable Data | -2.67 (2.89) | -2.00 (3.46)

ADVERSE EVENTS:
Time Frame: Up to one month
Groups:
- Burst-SCS: Participants received burst spinal cord stimulation (Burst-SCS), a neuromodulation therapy that delivers patterned electrical pulses in bursts to the spinal cord to help manage chronic pain. Burst-SCS aims to mimic natural neuronal firing patterns and may provide pain relief with reduced paresthesia. Stimulation was delivered using the St. Jude Medical Invisible Trial System. Study evaluations were conducted both before and after the intervention.
- Sham-SCS: Participants in this group received sham spinal cord stimulation (Sham-SCS), a control condition in which the stimulation device was programmed but the output amplitude was set to 0 mA, so no electrical stimulation was delivered. This approach mimics device use without activating the therapeutic effect, serving as a placebo control for the study. The St. Jude Medical Invisible Trial System was used for all procedures. Study evaluations were conducted both before and after the intervention.
Arm/Group | Burst-SCS | Sham-SCS
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/25/NCT03718325/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT03718325/ICF_001.pdf